CLINICAL TRIAL: NCT04728451
Title: Spectacle Prescribing in Early Childhood (SPEC)
Brief Title: Spectacle Prescribing in Early Childhood
Acronym: SPEC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Dan Twelker, Professor, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1911187060; UG1EY029657 (NIH)
Record Dates: First submitted 2021-01-21; First posted 2021-01-28 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Astigmatism Bilateral; Eyeglasses
Keywords: Astigmatism; Infant; Child, Preschool; Cognitive Development; Motor Development; Language Development; Child Development; Visual Acuity
MeSH Terms: conditions — Astigmatism | interventions — Eyeglasses

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full-Time Spectacle Wear (Active Comparator): Parents are asked to encourage their child to wear the spectacles full-time (all waking hours). A study staff member works closely with families throughout the child's participation to provide support and encouragement and to make suggestions on methods parents can use to maximize spectacle wear.
  Interventions: Behavioral: Spectacle wear support; Device: Spectacles
- Ad-Lib Spectacle Wear (Active Comparator): Parents are asked to encourage their child to wear the spectacles as much as possible for the initial 30 days after dispensing, and thereafter to continue to offer the spectacles to the child but not force the child to wear them if they resist or refuse. Limited support for parents is provided with regard to maximizing spectacle wear.
  Interventions: Device: Spectacles

INTERVENTIONS:
Behavioral: Spectacle wear support — Parents of children in the full-time group are provided with encouragement, support, and counseling throughout the study in order to maximize their child's spectacle wear.
  Arms: Full-Time Spectacle Wear
Device: Spectacles — Children prescribed and provided spectacles with full correction of their refractive error, with the exception of prescriptions with ≥ +1.50D sphere (plus cylinder notation) in the least hyperopic eye, which will be symmetrically reduced by 1.00D

SUMMARY:
The purpose of this study is to compare developmental outcome for young children (12 to 35 months of age) with astigmatism meeting American Academy of Ophthalmology spectacle prescribing guidelines and who are prescribed and provided spectacles for either Full-Time wear (encouraged and reinforced) or Ad Lib wear (wear dependent on child acceptance).

DETAILED DESCRIPTION:
The benefits and drawbacks of spectacle treatment for bilateral astigmatism in young children are not known. The SPEC study compares outcomes for young children (12 to < 35 months of age) with astigmatism meeting spectacle prescribing recommendations and randomized to either Full-Time spectacle wear (encouraged and reinforced) or Ad Lib spectacle wear (only as accepted by the child). The primary outcome analysis compares cognitive development at 38-42 months in children randomized to the Full-Time and Ad Lib groups. Secondary analyses compare Language, Motor, Social-Emotional, and Adaptive Behavior developmental outcomes and visual acuity outcome for children randomized to the Full-Time and Ad Lib groups.

ELIGIBILITY:
Inclusion Criteria:

* Parent/guardian provision of signed and dated informed consent form for Baseline/Eligibility Examination.
* Completion of Baseline/Eligibility Examination with cycloplegia.
* Bilateral astigmatism: Astigmatism ≥2.25D in the most astigmatic eye and ≥1.75D in the fellow eye based on manual cycloplegic retinoscopy conducted at Baseline/Eligibility Examination.
* Parent/guardian willing to accept assignment to either randomized group.
* Parent/guardian provision of signed and dated informed consent form for randomized SPEC Study.
* Parent willing to commit to study visits every 180 days, to be contacted (phone, email, or text) for reports of spectacle wear, and to allow their child to wear the TheraMon® sensor on the spectacle headband.
* Child and Family are primarily English or Spanish speaking.
* Parent/guardian does not anticipate moving out of Tucson area prior to their child reaching age 1275 days (approximately age 3 ½ years).
* Parent/guardian has not enrolled another child in the SPEC trial.

Exclusion Criteria:

* Gestational age <32 weeks (per parent report).
* Anisometropia ≥1.50 D spherical equivalent per manual cycloplegic retinoscopy conducted at the Baseline/Eligibility Examination.
* Current manifest strabismus per Baseline/Eligibility Examination.
* Ocular pathology per Baseline/Eligibility Examination (H44* or H25* diagnosis code).
* Previously diagnosed manifest strabismus or other ocular abnormalities (per parent report and per medical record):

  * H25* (Cataract)
  * H44* (Disorders of the Globe)
  * H50* (Strabismus)
  * H55* (Irregular Eye Movement and Nystagmus)
  * Q15.0 (Congenital Glaucoma)
  * Other diagnosis of an ocular abnormality
* Previous spectacle wear, amblyopia therapy, or vision therapy (per parent report and per medical record).

  * H53* (Amblyopia)
  * Other spectacle wear, amblyopia therapy, or vision therapy
* Current or previous diagnosis of developmental or neurological conditions (per parent report and per medical record):

  * H90.5 Congenital Deafness, and related disorders of hearing loss.
  * G40.909 Epilepsy or other seizure disorder.
  * P07.34 Prematurity 31 weeks, and other prematurity less than 32 weeks.
  * P91.6 Hypoxic Ischemic Encephalopathy
  * Q90.9 Down Syndrome, and other congenital syndromes associated with developmental delay.
  * Q04.4 Septo-Optic Dysplasia
  * Q91-Q92 Trisomy Other (13, 18, partial, complete, unbalanced translocations, mosaicism, duplications)
  * R62.50 Developmental Delay, and related disorders exhibiting a delay in one or more streams of development (e.g. language, fine motor, gross motor, social).
  * Other diagnosis of a developmental or neurological condition
* History of allergic response to dilating eye drops (per parent report):

  * Local redness and swelling of the eyelid consistent with contact dermatitis which resulted in the parent being informed that the child had a drug allergy to one of the dilating eye drops (proparacaine or cyclopentolate) or one of the carrier or preservative agents used in the formulation of these drops.

Ages: 12 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 88 (Estimated)
Dates: Start 2021-03-25 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Cognitive Development | Measured at the Developmental and Visual Assessment Visit (when the child is age 1155-1275 days)
  Cognitive Scale Composite Score on the "Bayley Scales of Infant and Toddler Development, 3rd Edition". Tester is masked to the child's randomized group. Scores (continuous scale) are based on published age norms (mean =100, standard deviation = 15) and range from 40-160 with higher scores indicating better outcomes. A difference of ≥10 points between randomized groups will be considered clinically meaningful.

SECONDARY OUTCOMES:
Language Development | Measured at the Developmental and Visual Assessment Visit (when the child is age 1155-1275 days)
  Language Scale Composite Score on the "Bayley Scales of Infant and Toddler Development, 3rd Edition". Tester is masked to the child's randomized group. Scores (continuous scale) are based on published age norms (mean =100, standard deviation = 15) and range from 40-160 with higher scores indicating better outcomes. A difference of ≥10 points between randomized groups will be considered clinically meaningful.
Motor Development | Measured at the Developmental and Visual Assessment Visit (when the child is age 1155-1275 days)
  Motor Scale Composite Score on the "Bayley Scales of Infant and Toddler Development, 3rd Edition". Tester is masked to the child's randomized group. Scores (continuous scale) are based on published age norms (mean =100, standard deviation = 15) and range from 40-160 with higher scores indicating better outcomes. A difference of ≥10 points between randomized groups will be considered clinically meaningful.
Social-Emotional Development | Measured at the Developmental and Visual Assessment Visit (when the child is age 1155-1275 days)
  Social-Emotional Scale Composite Score on the "Bayley Scales of Infant and Toddler Development, 3rd Edition". Tester is masked to the child's randomized group. Scores (continuous scale) are based on published age norms (mean =100, standard deviation = 15) and range from 40-160 with higher scores indicating better outcomes. A difference of ≥10 points between randomized groups will be considered clinically meaningful.
Adaptive Behavior | Measured at the Developmental and Visual Assessment Visit (when the child is age 1155-1275 days)
  Adaptive Behavior Scale Composite Score on the "Bayley Scales of Infant and Toddler Development, 3rd Edition". Tester is masked to the child's randomized group. Scores (continuous scale) are based on published age norms (mean =100, standard deviation = 15) and range from 40-160 with higher scores indicating better outcomes. A difference of ≥10 points between randomized groups will be considered clinically meaningful.
Visual Acuity | Measured at the Developmental and Visual Assessment Visit (when the child is age 1155-1275 days)
  Binocular visual acuity tested using the Amblyopia Treatment Study HOTV Protocol. Child wears most recent prescription for testing (or no spectacles, if discontinued by study doctor). Tester is masked to the child's randomized group. Acuity is recorded and analyzed as log MAR values (continuous scale). A difference of 0.10 log MAR between randomized groups will be considered clinically meaningful.

OTHER OUTCOMES:
Duration of spectacle wear | From the date of dispensing of the first pair of spectacles at the Spectacle Prescription Verification Visit through the date of the Developmental and Visual Assessment Visit, up to 30 months.
  Objective measures of duration of spectacle wear (hours/day) assessed objectively with a TheraMon® sensor attached to the child's spectacles. Temperature samples are recorded by the sensor every 15 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Erin M Harvey, Ph.D., Principal Investigator — University of Arizona; John D Twelker, O.D., Ph.D., Principal Investigator — University of Arizona
Locations (1):
- The University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Data Sharing Policy and Policy on the Dissemination of NIH-Funded Clinical Trial Information and the Clinical Trials Registration and Results Information Submission rule. De-identified data will be available upon request after publication by contacting the study Principal Investigators.
Supporting Information: Study Protocol, ICF
Time Frame: De-identified data will be available upon request after publication.
Access Criteria: De-identified data will be available upon request after publication by contacting the study Principal Investigators.